CLINICAL TRIAL: NCT04830930
Title: A Randomized, Open-label, Single-dose, Crossover Study to Investigate the Effect of Food on the Pharmacokinetics and Pharmacodynamics of CKD-381 in Healthy Volunteers
Brief Title: A Study to Investigate the Effect of Food on the PK, PD of CKD-381 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A73_04FDI2102
Record Dates: First submitted 2021-04-01; First posted 2021-04-05 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-03

CONDITIONS: GERD
Keywords: CKD-381
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Intervention Model Description: Crossover Assignment
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence 1 (Experimental): Period 1: fasted condition/ Period 2: fed condition
  Interventions: Drug: CKD-381
- Sequence 2 (Experimental): Period 1: fed condition/ Period 2: fasted condition
  Interventions: Drug: CKD-381

INTERVENTIONS:
Drug: CKD-381 — single-dose, oral administration of CKD-381 1 tablet

SUMMARY:
A study to investigate the effect of food on the Pharmacokinetics and pharmacodynamics of CKD-381 in healthy volunteers

DETAILED DESCRIPTION:
A randomized, open-label, single-dose, crossover study to investigate the effect of food on the pharmacokinetics and pharmacodynamics of CKD-381 in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Between 19 aged and 50 aged in healthy adult
2. Body weight more than 55.0kg and body mass index over 18.0kg/m2 and under 30.0kg/m2
3. Have negative result on Helicobacter Pylori antibody test

Exclusion Criteria:

1. Have clinically significant disease that hepatobiliary system, kidney, nervous system, immune system, respiratory system, endocrine system, hemato-oncology disease, cardiovascular system or mental illness, or a history of mental disease.
2. Have a gastrointestinal disease history(including surgery) that can effect evaluation of safety, pharmacokinetics and pharmacodynamics of investigational product.
3. Hypersensitivity reaction or clinically significant hypersensitivity reaction in the history of investigational product, additives or benzimidazole family.

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2021-04-21 (Actual); Primary Completion 2021-06-17 (Actual); Study Completion 2021-07-26 (Actual)

PRIMARY OUTCOMES:
Cmax | 0-24 hours
  maximum observed concentration after dose
AUClast | 0-24 hours
  Area under the plasma concentration versus time curve over the dosing interval after dose
Percent decrease from baseline in integrated gastric acidity for 24-hour interval after dose | 0-24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Kyungsang Yu, M.D., Ph.D., Principal Investigator — ksyu@snu.ac.kr
Locations (1):
- Seoul National University Hospital, Seoul, Jongno-gu, South Korea

IPD SHARING:
Plan to Share IPD: No